CLINICAL TRIAL: NCT07300917
Title: Efficacy and Safety of a 1726-nm Sebaceous-Targeting Diode Laser for the Treatment of Fordyce Spots of the Lips: A Prospective Pilot Study
Brief Title: 1726-nm Diode Laser for Lip Fordyce Spots
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Research Center (Other)
Responsible Party: Principal Investigator, Mahmoud Rageh, Dermatologist, Venus Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Accure_Fordyce_Spots
Record Dates: First submitted 2025-12-21; First posted 2025-12-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Fordyce Spots
Keywords: Fordyce spots; Sebaceous glands; Lip lesions; Cosmetic dermatology; Diode laser; 1726 nm laser
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Accure 1726-nm Laser Treatment (Experimental): Participants receive treatment to the entire affected lip and/or vermilion area using a 1726-nm sebaceous-targeting diode laser (Accure®) delivered in 2-3 sessions at four-week intervals.
  Interventions: Device: Accure 1726-nm Diode Laser

INTERVENTIONS:
Device: Accure 1726-nm Diode Laser — A 1726-nm sebaceous-targeting diode laser (Accure®) delivering multi-pulse, temperature-guided energy with continuous cooling, applied to the lips and vermilion border in 2-3 treatment sessions spaced four weeks apart.

SUMMARY:
Fordyce spots are benign ectopic sebaceous glands commonly affecting the lips and vermilion border, often causing cosmetic concern. This prospective pilot study evaluates the efficacy and safety of a 1726-nm sebaceous-targeting diode laser (Accure®) for the cosmetic treatment of Fordyce spots of the lips. Participants will receive 2-3 laser sessions and will be followed for 6-12 months to assess clinical improvement, patient satisfaction, and safety outcomes.

DETAILED DESCRIPTION:
This is a prospective, single-arm pilot study evaluating the use of a 1726-nm diode laser that selectively targets sebaceous glands via lipid absorption. The device employs a temperature-guided, multi-pulse delivery system with continuous cooling and is FDA-cleared for the treatment of inflammatory acne.

Eligible participants with clinically evident Fordyce spots of the lips and/or vermilion border will receive 2-3 treatment sessions spaced four weeks apart. Outcomes include lesion count reduction, global aesthetic improvement scores, patient satisfaction, and safety assessments. Follow-up visits will occur at Weeks 4, 8, 12, 24. To better characterize durability and recurrence, participants will be invited (optional) to return for an additional observational follow-up at Month 12 (±4 weeks), without any additional study treatment. Participants who do not attend the Month-12 visit will be considered complete after the Week-24 assessment and will not be contacted further beyond routine clinical care. All analyses of efficacy and safety will be based on assessments through Week 24, with Month-12 data summarized descriptively as extended follow-up where available.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinically evident Fordyce spots involving: Upper and/or lower lips and/or vermilion border
* Cosmetic concern related to Fordyce spots
* Willingness to comply with study procedures and follow-up visits
* Ability to provide written informed consent

Exclusion Criteria:

* Active herpes labialis at the treatment site
* History of frequent HSV reactivation without willingness for antiviral prophylaxis
* Isotretinoin use within the preceding 6 months
* Active inflammatory or infectious lip/mucosal disease (e.g., lichen planus, cheilitis, candidiasis)
* Known tendency for keloid or hypertrophic scarring Pregnancy or lactation
* Immunosuppression or uncontrolled systemic illness
* Previous treatment of Fordyce spots in the target area within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage Reduction in Fordyce Spot Count | Baseline to Week 12
  The percentage change from baseline in the number of visible Fordyce spots on the lips and vermilion border, assessed using standardized clinical photographs and lesion counting within predefined grid areas.

SECONDARY OUTCOMES:
Investigator Global Improvement Assessment (IGA) | Baseline to Week 12
  Change in investigator-rated global improvement using a 5-point scale ranging from no improvement to almost complete clearance.
Patient Global Aesthetic Improvement Scale (Patient-GAIS) | Baseline to Week 12
  Patient-reported global aesthetic improvement assessed using a 5-point scale ranging from no improvement to almost complete clearance.
Patient Satisfaction Score | Week 12
  Patient satisfaction with cosmetic outcome assessed using a visual analog scale from 0 (not satisfied) to 10 (extremely satisfied).
Treatment Safety and Tolerability | Baseline to Month 6
  Incidence and severity of treatment-related adverse events including pain, erythema, edema, mucosal erosion, ulceration, pigmentary changes, and herpes labialis reactivation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hosn Clinics, Khobar, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including baseline characteristics, lesion counts, and outcome measures, will be shared.
Time Frame: Beginning 6 months after publication and available for 5 years.
Access Criteria: Data will be shared upon reasonable request to the corresponding author, following approval of a methodologically sound proposal and execution of a data use agreement.